CLINICAL TRIAL: NCT07042373
Title: Innovative Policy: Effects of Tobacco Abuse Liability-dependent Taxes in the ETM
Brief Title: Effects of Tobacco Abuse Liability-dependent Taxes in the ETM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: VT IRB # 23-729; 5K01CA279490-02 (NIH)
Record Dates: First submitted 2025-05-27; First posted 2025-06-29 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-05

CONDITIONS: Cigarette Smoking Behavior
Keywords: Cigarettes; Experimental Tobacco Marketplace; Abuse Liability
MeSH Terms: conditions — Cigarette Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cigarette smokers (Experimental): In a within-subject design, cigarette smokers, stratified by age, will purchase tobacco products under three tax rate conditions based on abuse liability, that is taxes based on: (1) product category score (i.e. score ranging from 0-1 based on abuse liability effect sizes); (2) product category rank (i.e. position of a product relative to all others; e.g. 1st, 5th); and (3) product tiers (i.e. low-, medium-, high abuse liability), as well as a control. In the ETM, the effects of these interventions will be examined on cigarette demand and other products substitution.
  Interventions: Behavioral: Control; Behavioral: Product Category Score; Behavioral: Product Category Rank; Behavioral: Product Tiers

INTERVENTIONS:
Behavioral: Control — In the control condition, participants will purchase tobacco/nicotine products in the ETM. Cigarettes will increase in price across trials.
Behavioral: Product Category Score — In the product category score condition, participants will purchase tobacco/nicotine products in the ETM where the percentage of taxes applied to each product category will be distributed between 0% and 100% proportional to their abuse liability score. Abuse liability scores will be scaled such that the product category with the highest abuse liability will be taxed at 100%.
Behavioral: Product Category Rank — In the product category rank condition, participants will purchase tobacco/nicotine products in the ETM where the tax percentage applied to each product category will be determined by the number of categories and their position in the ranking. The product category with the highest abuse liability will be taxed at 100%; the product with the lowest abuse liability will be taxed at 0%. All other tax rates will be equally spaced across other products based on ranking.
Behavioral: Product Tiers — In the product tiers condition, participants will purchase tobacco/nicotine products in the ETM where tobacco products will be placed in tax tiers to simplify the existing complex tobacco tax system. The investigators will use three tax tiers (i.e., high tax, medium tax, and no tax), as adopted by four states. Products will be placed into tiers depending on their average score (i.e. no tax: < 0.33, medium tax: 0.33-0.66, and high tax: >0.66). Products in the high tax tier will be taxed at 100% and products in the medium tax tier will be taxed at 50%.

SUMMARY:
In a within-subject design, cigarette smokers, stratified by age, will purchase tobacco products under three tax rate conditions based on abuse liability, that is taxes based on: (1) product category score (i.e. score ranging from 0-1 based on abuse liability effect sizes); (2) product category rank (i.e. position of a product relative to all others; e.g. 1st, 5th); and (3) product tiers (i.e. low-, medium-, high abuse liability), as well as a control. In the ETM, the effects of these interventions will be examined on cigarette demand and other products substitution.

The investigators will use a repeated-measures (within subject) analysis of variance (ANOVA) to test if there are differences between conditions (i.e., tax proposals) independently for each product. The models will include study design parameters for order effects to account for counterbalancing the tax conditions in the ETM. Each tax condition will be compared to the control. All distributional assumptions will be checked prior to analyses and the appropriate transformations will be employed, if needed. For each significant result from the omnibus test, the investigators will perform planned contrasts to test the proposed hypotheses previously described. Note that the omnibus test can result in a significant finding while the contrasts of interest may be non-significant. In this case, the investigators will only report the results from the planned contrasts.

Additional analyses might be conducted.

DETAILED DESCRIPTION:
In this study, the investigators will experimentally examine the impact of abuse-liability taxes on tobacco product purchases and ultimately tobacco dependence.

The investigators hypothesize that (1) the three abuse-liability tax proposals (product category score; product category rank; product tiers) will decrease purchasing of products with the highest abuse liability; and (2) increase purchasing of products with lower abuse liability (substitution) compared to control. Moreover, (3) the tax rate based on product category score will lead to the greatest substitution, because it is most reflective of abuse liability differences.

In a within-subject design, cigarette smokers stratified by age will complete one control trial and three ETM conditions representing the three tax rates based on abuse liability. Within each condition, taxes will be increased proportionally across 5 trials to examine how cigarette purchasing and substitution are affected.

The study will consist of two in-lab visits and one phone call visit: 1) a consent and assessments session 2) an ETM session, and a 3) follow-up phone-call session approximately 7 days after session 2. Session 1 and 2 will be separated by an at home product sampling phase.

1. Session 1: Consent and Assessments In the consent and initial assessment session, participants will go through standard consent procedures. Participants will provide a breath sample to confirm recent levels of smoking that will be measured using a CoVita® Micro+ Basic Smokelizer. Women of child-bearing age will provide a urine sample to test for pregnancy. Participants will complete a timeline follow back to assess previous month smoking habits and consumption of nicotine products to determine ETM budget. Participants will complete a survey with demographic questions and nicotine/tobacco-related assessments (Fagerstrom Test for Cigarette Dependence, Perceived Health Risk adapted, Questionnaire on Smoking Urges-Brief, Motivation to Quit, Self-efficacy to Quit, and The Contemplation Ladder adapted).

   For the at home sampling period, participants will be shown a menu of the products available for purchase in the ETM. Participants will choose one product from each category, to sample at home, before the next session (approximately 4 days later). Participants will receive instructions to use the products over the next four days. Participants will complete a product evaluation scale for each product. Participants will be asked if they sampled each product as instructed.
2. Session 2: ETM In the ETM session, participants will be provided with an individual 7-day experimental budget calculated based on their average tobacco/nicotine consumption over the past 30 days. For example, if a participant reports smoking 20 cigarettes per day (a pack), they will receive $35.00, equivalent to 140 cigarettes (or 7 packs) multiplied by $0.25 per cigarette (market price of an individual cigarette) to spend in the ETM. In the ETM, first, participants will experience two practice trials. Then, participants will complete the real ETM consisting of one control trial and three tax rate conditions based on abuse liability. Conditions will be balanced in a latin square design to account for any other effects. Participants will complete a total of 20 purchasing trials each for 7 days worth of products. In each trial, participants will buy tobacco products to use throughout the next 7 days. At the end of the session, the participant will randomly draw an individual purchasing trial and will receive all the products purchased at that trial to use over the next week. During the following 7 days, the participant is asked to use only the tobacco/nicotine products received during the study.
3. Session 3: Follow-up In the follow-up session, participants will receive a phone call from study personnel who will complete a timeline follow back interview to assess previous week recent smoking, and consumption of nicotine products, Product Evaluation Scale, Motivation to Quit, Self-efficacy to quit, The Contemplation Ladder adapted, and Experiment/Experimenter Attitudes Rating Scale. These questions may be asked over the phone and/or using zoom.

ELIGIBILITY:
Inclusion criteria:

* Provide informed consent
* Be at least 21 years of age or older
* Provide a breath sample for measuring carbon monoxide (CO ≥ 8 ppm)
* Smoke at least 10 cigarettes daily
* Use other tobacco products less than weekly

Exclusion criteria:

* Have uncontrolled physical or mental health conditions
* Use of smoking cessation medications (e.g., nicotine replacement, bupropion, varenicline) in the past 30 days
* Report concrete, immediate plans to alter/quit using their usual tobacco products in the next 30 days
* If they are pregnant or lactating
* Have plans to move out of the area during the experiment

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Cigarette Demand Intensity | Day 1
  Participants will complete purchasing trials in an Experimental Tobacco Marketplace (ETM), where nicotine/tobacco prices will increase accordingly with the condition. The quantity of products purchased in the ETM will be converted to milligrams (mg) of nicotine to standardize the unit of measurement across products. The data will reflect the relationship between nicotine purchased (mg; y-axis) and cigarette price (x-axis). Demand will be estimated using the exponential equation: Q = Q0 * 10^k(exp(-αQ0C) - 1), where Q is nicotine purchased (mg), C is price, Q0 is demand intensity (purchases at no cost), k is the function's logarithmic span, and α is demand elasticity. Intensity will be reported, which represents the estimated mg of nicotine purchased when cigarettes are free (price = 0).
Cigarette Demand Elasticity | Day 1
  Participants will complete purchasing trials in an Experimental Tobacco Marketplace (ETM), where nicotine/tobacco prices will increase accordingly with the condition. The quantity of products purchased in the ETM will be converted to milligrams (mg) of nicotine to standardize the unit of measurement across products. The data will reflect the relationship between nicotine purchased (mg; y-axis) and cigarette price (x-axis). Demand will be estimated using the exponential equation: Q = Q0 * 10^k(exp(-αQ0C) - 1), where Q is nicotine purchased (mg), C is price, Q0 is demand intensity (purchases at no cost), k is the function's logarithmic span, and α is demand elasticity. Elasticity will be reported, which represents the sensitivity of purchasing to changes in cigarette price.
Nicotine/Tobacco Products Substitution Slope | Day 1
  Participants will complete purchasing trials in an Experimental Tobacco Marketplace (ETM), where nicotine/tobacco prices will increase accordingly with the condition. The quantity of products purchased in the ETM will be converted to milligrams (mg) of nicotine to standardize the unit of measurement across products. The data will reflect the relationship between nicotine purchased (mg; y-axis) and cigarette price (x-axis).
  To obtain estimates of substitution of price-constant products in the different ETM conditions, the investigators will use ordinary least squares regression to predict total mg of nicotine purchased of the price-constant product. Slope of price-constant products will be reported, which represents the change in mg of nicotine purchased of price-constant products divided by the change in cigarette price.
Nicotine/Tobacco Products Substitution Intercept | Day 1
  Participants will complete purchasing trials in an Experimental Tobacco Marketplace (ETM), where nicotine/tobacco prices will increase accordingly with the condition. The quantity of products purchased in the ETM will be converted to milligrams (mg) of nicotine to standardize the unit of measurement across products. The data will reflect the relationship between nicotine purchased (mg; y-axis) and cigarette price (x-axis). To obtain estimates of substitution of price-constant products in the different ETM conditions, the investigators will use ordinary least squares regression to predict total mg of nicotine purchased of the price-constant product. Y-intercept of price-constant products will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Roberta Freitas Lemos, Ph.D., Principal Investigator — Fralin Biomedical Research Institute at VTC
Locations (1):
- Fralin Biomedical Research Institute at VTC, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Demographical, behavioral, and ETM data will be stored within a secure computing environment. All direct respondent identifiers (e.g., names and addresses) will be removed and maintained in a secure file for future contact purposes. Data from this project will be preserved to enable sharing via NDA with sufficient quality to validate and replicate research findings. All data will be provided in .CSV format. Respondent identifiers will not be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The research community will have access to data upon publication of this study, consistent with the NDA guidelines. NDA will make decisions about how long to preserve the data.
Access Criteria: Researchers will use the standard processes at NDA to request access to the data. The NDA Data Access Committee will decide which requests to grant. The standard NDA data access process allows access for one year and is renewable.

REFERENCES:
- [Background] Chaloupka FJ, Grossman M, Bickel WK, Saffer H. The Economic Analysis of Substance Use and Abuse: An Integration of Econometric and Behavioral Economic Research. 1999 Jan 1
- [Background] Freitas-Lemos R, Keith DR, Tegge AN, Stein JS, Cummings KM, Bickel WK. Estimating the Impact of Tobacco Parity and Harm Reduction Tax Proposals Using the Experimental Tobacco Marketplace. Int J Environ Res Public Health. 2021 Jul 23;18(15):7835. doi: 10.3390/ijerph18157835. PMID 34360124
- [Background] Stiles MF, Campbell LR, Graff DW, Jones BA, Fant RV, Henningfield JE. Pharmacodynamic and pharmacokinetic assessment of electronic cigarettes, combustible cigarettes, and nicotine gum: implications for abuse liability. Psychopharmacology (Berl). 2017 Sep;234(17):2643-2655. doi: 10.1007/s00213-017-4665-y. Epub 2017 Jun 20. PMID 28634710
- [Background] Shakhnovich V. It's Time to Reverse our Thinking: The Reverse Translation Research Paradigm. Clin Transl Sci. 2018 Mar;11(2):98-99. doi: 10.1111/cts.12538. Epub 2018 Feb 9. No abstract available. PMID 29423973
- [Background] Pope DA, Poe L, Stein JS, Kaplan BA, DeHart WB, Mellis AM, Heckman BW, Epstein LH, Chaloupka FJ, Bickel WK. The Experimental Tobacco Marketplace: Demand and Substitutability as a Function of Cigarette Taxes and e-Liquid Subsidies. Nicotine Tob Res. 2020 Apr 21;22(5):782-790. doi: 10.1093/ntr/ntz116. PMID 31350894